CLINICAL TRIAL: NCT00814021
Title: Phase II Study, Multicenter, Open-label, Evaluating Efficacy of Treatment With Sutent® (Sunitinib) in Patients With Previously Untreated or Recurrent Brain Metastases Originating From Renal Cancer
Brief Title: Sunitinib in Treating Patients With Kidney Cancer That Has Spread to the Brain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07URO02; ICREGAUD-07URO02; ICREGAUD-Metastases Cerebrales; INCA-RECF0821; PFIZER-ICREGAUD-07URO02; EUDRACT-2008-000948-13
Record Dates: First submitted 2008-12-20; First posted 2008-12-23 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2012-08

CONDITIONS: Kidney Cancer; Metastatic Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; tumors metastatic to brain
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell; Brain Neoplasms | interventions — Sunitinib

ARMS (1):
- sunitinib, (Experimental)
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with kidney cancer that has spread to the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in the brain after 2 courses of sunitnib malate in patients with previously untreated or recurrent brain metastases secondary to renal cancer following radiotherapy or surgery.

Secondary

* Evaluate duration of response.
* Evaluate objective response of non-CNS targets.
* Evaluate time to disease progression.
* Evaluate overall and progression-free survival.
* Evaluate neurological symptoms associated with the tumor.
* Evaluate feasibility and overall tolerance of this drug.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the kidney

  * Metastatic disease
* Measurable disease by RECIST criteria
* Presence of previously untreated or recurrent brain metastases following radiotherapy or surgery

  * No brain metastasis revealed by hemorrhage
  * No single brain metastasis < 2 cm that is accessible by surgery or radiosurgery

PATIENT CHARACTERISTICS:

* WHO performance status 0-2 (unless paresis due to brain metastases)
* ANC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8 g/dL
* PT or INR < 1.5 times upper limit of normal (ULN)
* AST/ALT < 2.5 times ULN (< 5 times ULN in the case of liver metastases)
* Total bilirubin < 1.5 times ULN
* Serum creatinine < 200 μmol/L
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for up to 30 days following completion of study treatment
* No other cancer except for in situ cervical cancer, curatively treated basal cell carcinoma of the skin, or other curatively treated cancer without evidence of recurrence within the past 5 years
* No uncontrolled hypertension (systolic BP ≥ 160 mm Hg and/or diastolic BP ≥ 90 mm Hg)
* None of the following cardiac conditions within the past 6 months:

  * Significant cardiovascular disease
  * NYHA class III-IV congestive heart failure
  * Myocardial infarction
  * Unstable angina
  * Severe arrhythmia
  * Cerebrovascular accident
  * Severe thromboembolism
* No serious neuropsychiatric disease
* No psychological, familial, social, or geographic situations that preclude clinical follow-up
* No patient deprived of liberty by a court or administrative order
* Able to understand French

PRIOR CONCURRENT THERAPY:

* At least 6 months since prior antineoplastic treatment with sunitinib malate
* At least 4 weeks since other prior treatment
* At least 3 weeks since prior hematopoietic growth factors (i.e., filgrastim [G-CSF] or sargramostim [GM-CSF])
* No concurrent antivitamin K at curative or anticoagulation doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate in the brain after 2 courses | From beginning of treatment until 2 courses of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chevreau-Dalbianco, MD, Study Chair — Institut Claudius Regaud
Locations (1):
- Institut Claudius Regaud, Toulouse, France